CLINICAL TRIAL: NCT02690428
Title: To Evaluate the Safety & Palliative Treatment Effect on Patients With Solid Cancers by Immunostimulating Interstitial Laser Thermotherapy (imILT)
Brief Title: Immunostimulating Interstitial Laser Thermotherapy in Solid Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient recruitment slow
Sponsor: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2014-003
Record Dates: First submitted 2016-02-15; First posted 2016-02-24 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Neoplasms
Keywords: Hyperthermia, Induced; Laser Coagulation; Laser Therapy
MeSH Terms: conditions — Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imILT (Experimental): Immunostimulating Interstitial Laser Thermotherapy (imILT)
  Interventions: Device: Immunostimulating Interstitial Laser Thermotherapy

INTERVENTIONS:
Device: Immunostimulating Interstitial Laser Thermotherapy — Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response.

SUMMARY:
Thermotherapy is a technology aiming at destroying tissue, for example tumor tissue. Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response. In laboratory animals the imILT method has also been shown to induce a so called abscopal effect. This means that when one tumor is treated with imILT other, untreated, tumors also decrease in size. The immunologic response has previously been characterized in breast cancer patients after receiving imILT treatment , and presumed abscopal effects induced by imILT have also been described in a malignant melanoma patient.

The purpose of this trial is to evaluate efficiency when it comes to local tumor destruction of the imILT treatment method in patients diagnosed with solid tumors. The purpose is also to investigate the functionality and safety as well as understanding of the subsequent immunological effects. Since immunologically based treatment of various solid tumors is under intense review with so called "immune checkpoint inhibitors" this trial will also provide valuable information on how imILT, in the future, could be combined with these new and, for some patients, very effective treatment regimens.

The treatment method has successfully been used for treatment of patients with breast cancer and malignant melanoma. Treatment of breast cancer patients caused an increase of cytotoxic T lymphocytes in the treated tumor, as well as activated dendritic cells at the tumor border. Regulatory T lymphocytes decreased in the regional lymph nodes.

This trial is explorative, prospective, open and non-randomized. Thirty patients diagnosed with solid tumors will be treated in this trial, which is estimated to be carried out during a time period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female > 18 years of age
* Have histologically confirmed, locally uncontrolled, solid cancer, with or without metastases, that cannot be treated surgically due to unresectability or inoperability
* Have one or more tumours assessable by MRI/CT or ultrasound and situated in such a way that at least a part of the tumour can be treated with IMILT without damage to surrounding vital structures or the skin
* Are candidates for ablative intervention also outside this study
* Have given informed verbal and written consent to participation in the trial
* Have an ECOG performance status < 2 (Karnofsky > 60%)
* Have stable haematologic, renal and hepatic functions

Exclusion Criteria:

* Are HIV positive
* Have an active autoimmune disease
* Are on systemic corticosteroid medication (local treatment with aerosol's and ointment is allowed)
* Have known bleeding disorders or are treated with anticoagulant medication
* Are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Treatment effect (Measurement of tumor burden by irRC criteria) | 18 months
  Measurement of tumor burden by irRC criteria.

SECONDARY OUTCOMES:
Inflammatory response in tumor measured by quantification of inflammatory cell populations | 18 months
  Quantification of cellular infiltrate and activation markers by immunohistochemistry.
Inflammatory response in circulation measured by quantification of inflammatory cell populations | 18 months
  Quantification of cellular infiltrate and activation markers by flow cytometry.
Safety (adverse events) | 18 months
  Evaluation of adverse events.
Evaluation of pain (measured by VAS) | 18 months
  Evaluation of pain is performed using the visual analog scale (VAS).
Evaluation of Quality of Life (using a standardized questionnaire) | 18 months
  Evaluation of Quality of Life is evaluated using a standardized questionnaire (EORTC, general).
Usability of the device as evaluated by treatment logs | 18 months
  Evaluation of the laser system by analysis of treatment logs of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No